CLINICAL TRIAL: NCT06761235
Title: Vascular Age As a Key for a Team-based Approach to Manage Blood Pressure Bridging Community Pharmacists and Primary Health Care Physicians - the TOGETHER Trial
Brief Title: Knowledge of Vascular Age Contributes to Improve the Collaboration Between Community Pharmacies and Primary Health Care Physicians in Reducing Blood Pressure in Hypertensive Patients.
Acronym: TOGETHER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Enrique Rodilla (Other)
Collaborators: Health Research Fund of ISCIII Spain (Unknown); AIT Austrian Institute of Technology GmbH (Other); Institut et Haute Ecole de la SantÃ© la Source (Unknown); Instituto PolitÃ©cnico de Coimbra (Unknown); European Union (Other)
Responsible Party: Sponsor-Investigator, Enrique Rodilla, PhD, full Professor, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: FP-1533-ROD-SAL-2024-01; THCS: FP-1533 (Other: JTC 2023 - Healthcare of the Future)
Record Dates: First submitted 2024-11-17; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Hypertension and Cardiovascular Risk Factors
Keywords: hypertension; Arterial stiffness; estimated Pulse Wave Velocity; Community Pharmacies; Primary Care; Vascular Age; Team-based Approach
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: No other parties masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blood pressure arm (BP arm) (Placebo Comparator): Optimized standard treatment for hypertensive patients
  Interventions: Diagnostic Test: Standard BP intervention
- Early vascular aging arm (EVA arm) (Experimental): Optimized standard treatment for hypertensive patients plus information about individual vascular age assessed by brachial oscillometry
  Interventions: Diagnostic Test: EVA intervention

INTERVENTIONS:
Diagnostic Test: Standard BP intervention — Behavioral: lifestyle counseling will be given according to international guidelines to reduce blood pressure.
  Other Names: Ambulatory blood pressure monitoring to diagnose hypertension and educational sessions to empower hypertensive patients
  Arms: Blood pressure arm (BP arm)
Diagnostic Test: EVA intervention — Behavioral: lifestyle counseling will be given according to international guidelines to reduce blood pressure. In contrast to BP arm, EVA arm will additionally reciuve counseling about vascular age.
  Other Names: Ambulatory blood pressure monitoring to diagnose hypertension plus estimated vascular age by brachial oscillometry and educational sessions to empower hypertensive patients
  Arms: Early vascular aging arm (EVA arm)

SUMMARY:
Cardiovascular diseases are the main cause of death worldwide and elevated blood pressure (BP), called hypertension (HTN), is the principal and most frequent factor for suffering cardiovascular diseases. Recent studies show that approximately five out of 10 adults in Europe have increased BP or will develop HTN in their life-course. Unfortunately, screening programs for establishing the diagnosis of HTN do not exist. As a result, almost half of hypertensive patients do not know that their BP is elevated. Regarding the other half of subjects, who have been already diagnosed of HTN and are aware of their condition, up to 50% of them are not adequately controlled, although successful treatment of HTN is possible. There are several reasons explaining why at the end only one quarter of the hypertensive population achieves normal BP values. Firstly, there is a lack of patients´ adherence to the prescribed treatment. In other words, many patients do not take their pills as ordered, mostly because they do not realize the health risks associated with HTN, as elevated BP does not hurt nor lead to clinical symptoms. As a matter of fact, many hypertensive patients do not comply with their prescribed treatments. Secondly, the mere fact of prescribing drugs for reducing elevated BP is very often considered enough by the treating general practitioners, not having into account that the target blood pressure values are not achieved. This attitude is called therapeutic inertia. And thirdly, there is a lack of efficient communication between those specialized groups of health professionals, which are involved in the management of HTN, i.e. general practitioners and community pharmacies. In the context of high BP, the concept of early vascular aging (EVA), presented roughly 10 years ago, has been widely adopted since. The concept of vascular age generally refers to a way of expressing cardiovascular risk as an estimated age, considered useful for improving the understanding of cardiovascular risk in patients, especially in young patients, in whom standard information about health risks, such as the classical 10 year-risk derived from risk tables, is low and may transmit a false reassuring perception. "Your arteries are 15 years older then you" seems to make vascular age intuitively understood even by lay people. Vascular age has been shown to be easily estimated in community pharmacies in different countries and may contribute to increase HTN control.

The goal of this clinical trial is to learn if increasing awareness of the consequences of elevated blood pressure by estimating vascular age of hypertensive patients in community pharmacies, and thus, empowering them, firstly, improves compliance with scheduled visits with general practitioners and secondly, increases hypertension control as measured by ambulatory blood pressure measurements (ABPM).

The main questions it aims to answer are:

* Do hypertensive patients who know their vascular age comply better with scheduled visits to their general practitioners than hypertensive patients not aware of their vascular age?
* Does knowledge of vascular age improve the proportion of controlled HTN according to ABPM measurements after six months of state of the art treatment? Researchers will compare two groups of hypertensive patients.
* One half of the patients, the BP-arm, will receive usual educational sessions and standard, optimized advice.
* The so-called EVA-arm will get the same educational sessions and advice, but on top will be informed about their vascular age. After six months, ABPM will be repeated in both groups.
* The study will take place in Austria, Portugal and Spain.

Participants:

* Participants are pharmacy customers who volunteered to participate.
* To enter the study, BP must be > 140/90 mmHg in the pharmacy and > 130/80 mmHg in the first ABPM.
* Recruitment and estimation of vascular age will take place in community pharmacies.
* Treatment will be established by the general physicians according to best clinical practice.
* The study will end after six months with a second measurement of ambulatory BP.

DETAILED DESCRIPTION:
The five challenges in controlling high blood pressure Poor control of Hypertension and absence of sustained screening strategies Cardiovascular (CV) diseases represent the principal cause of death in Europe with 343.4 deaths/100,000 inhabitants, clearly ahead cancer with 235.3 deaths/100,000 inhabitants/year in 2021. Within the three different countries participating in TOGETHER, Austria (AT), Portugal (PT) and Spain (ES), AT ranks first with 343.3 CV deaths/100,000 inhabitants/year, followed by PT and ES, with 247.9 and 213.0 CV deaths/100.000 inhabitants/year, respectively1.

High blood pressure (BP), known as arterial hypertension (HTN), is the leading risk factor for CV diseases and hence for disability and mortality worldwide. According to a recent review of 12 western countries showed prevalence rates between 33% and 56%, knowledge rates between 46% and 84%, treatment rates between 39% and 81% and control rates between 17% and 69%.

Unfortunately, reliable data on prevalence and treatment of HTN in the three participating countries are scarce. In May 2017, as part of the International Society of Hypertension (ISH) "May Measurement Month"-campaign, standardized BP measurements were conducted in 80 countries around the world in various locations. In AT, 56 centers participated in the initiative and a total of 2,711 people were screened for HTN. Of these, 1,704 (62.9%) had BP values > 140/90 mmHg. Participants were also provided with comorbidities and medication assessment sheets, which showed that 43.2% of subjects without antihypertensive treatment were hypertensive. The result for people who were already taking antihypertensive therapy was particularly worrying as 63.5% had uncontrolled HTN.

The results of the same MMM-2017-campaign in ES were similar. 7,646 subjects participated throughout ES, 40.0% presented with HTN, of which 74.4% were aware of their disease, while up to 25.6% of patients with high BP levels were unaware of their HTN status. Among participants who were not taking antihypertensive drugs, elevated values were measured in 16.9%. Another worrying finding is that in treated hypertensive patients, 36.4% had not controlled values.

In PT, the prevalence of HTN in the adult population was estimated to be 42.2% in the PHYSA study, a representative sample of the 18-90-year-old population, including 3,720 participants, with 70% of the HTN patients under pharmacological medication. The age-specific prevalence of hypertension was 6.8, 46.9 and 74.9% in people below 35 years, 35-64 years and above 64 years, and overall, among the hypertensive patients, 76.6% were aware of the HTN condition, 74.9% were treated but only 42.5% were controlled.

Despite the enormous significance of HTN and the very low rates of control of elevated BP, there are currently no established population-screening programs aimed at diagnosing HTN in most countries around the world.

Deficiencies in estimating cardiovascular risk using risk tables The implementation of the concept of CV risk stratification in the late nineties of the last century has represented a significant milestone in the prevention of coronary and cerebrovascular diseases. The first risk tables were developed in the USA from five variables easy to determine, such as gender, age, smoking habit, systolic BP and LDL cholesterol. Subsequently, and with European population data, risk estimates were calculated in Europe that have finally been consolidated as reference tables, the so-called SCORE Tables. Its later development, following a very similar methodology and with only small differences, has resulted in SCORE2 and SCORE-OP (OP: old people) to integrate people over 65 years.

Nevertheless, the prognostic value of all known risk tables is limited in daily routine. Although the relative risk of an individual patient is much higher in the group of patients classified as high-risk compared to the other groups, it is equally indisputable that, in people in the same age group in absolute figures, more patients die in the group of patients classified as low or intermediate risk than in the group of high risk, as evidenced by a large number of studies, also in Middle-Europe. This is because there are many more patients in the low and moderate risk group than in the high and very high-risk group. To overcome this difficulty, in 1999 the concept of subclinical target organ damage (TOD) was introduced as a parameter that modifies the prognosis of patients independently and additively to the presence of CV risk factors. These are intermediate risk markers that can be diagnosed in asymptomatic patients usually before the appearance of established clinical diseases. The risk tables of the European Society of Hypertension (ESH) state that the mere presence of TOD in a patient, even with BP figures in the normal-high range, significantly modifies their CV risk. Avoiding the appearance of TOD, achieving its regression or at least delaying its progression is the strategy proposed by the ESH Guidelines, which recommend the determination of TOD whenever possible as an aid to the management of hypertensive patients.

Hypertension mediated organ damage (HMOD) may involve different organs, at the cardiac level, left ventricular hypertrophy, and at the renal level the increase in urinary albumin excretion and reduced glomerular filtration rate, both difficult to determine in large-scale HTN screening campaigns.

The third HMOD is located in the arterial system and involves different facets. The most widespread and known vascular HMOD is atherosclerosis, an alteration that mainly affects arterial lumen. A different HMOD is called arteriosclerosis or arterial stiffness, a condition in which mainly the arterial wall and pulse wave propagation characteristics are altered. Both terms, "atherosclerosis" and "arteriosclerosis", are frequently used in the literature as synonyms. And although they often overlap and share risk factors, these are different pathophysiological entities. Arteriosclerosis is mainly due to the replacement of elastin fibers by collagen of a more rigid nature and complex changes of muscle fibers in the media. These changes in the arterial wall produce an increase in PWV, evidencing increased arterial stiffness, as well as the development of isolated systolic HTN, elevated pulse pressure and accelerated (early) vascular aging (EVA). In contrast, in atherosclerosis, proinflammatory cells of the immune system, smooth muscle cells, lipids and connective tissue accumulate in the intima of arterial walls, reducing and obstructing arterial lumen. Even though both athero and arteriosclerosis express the cumulative exposure of aggressors to the arterial wall, arteriosclerosis tend to occur earlier in the CV continuum, therefore assessing arteriosclerosis might provide a more precocious indication of HTN mediated arterial wall damage. Atherosclerosis can be easily diagnosed by ultrasound of superficial arteries. Its availability is limited to specialized units and it cannot thus be recommended as a tool for large-scale population screening.

The gold standard method for assessing arteriosclerosis (arterial stiffness) is carotid-femoral applanation tonometry to measure PWV between the femoral artery and the carotid artery. It is a complex technique that requires training, time and equipment not currently affordable to perform a population-based screening. However, the AIT Austrian Institute of Technology (AIT, Vienna) and collaborators have developed and validated a new method for estimating aortic PWV from the pressure wave morphology, blood pressure and age in recent years, a simple and repeatedly validated technique allowing the estimation of the aortic PWV using the widely available method of brachial oscillometry. It consists technically of a procedure similar to a BP measurement that indirectly calculates arterial parameters in just a few minutes.

Validation studies, the establishment of normal values and extensive experience in various countries makes PWV estimation from brachial arterial BP cuffs a viable option for detecting subclinical vascular damage in large-scale clinical studies and clinical routine. Thus, in a large-scale comparative study with approximately 900 participants, estimation of PWV by non-invasive means by brachial oscillometry was found to be a feasible alternative to the exact determination of PWV by an invasive intra-arterial catheter. In fact, the standard deviation of the PWV estimation by oscillometry with respect to invasive measurement was lower than the standard deviation by means of the carotid-femoral tonometry mentioned above. Subsequently, another validation of the method was carried out against a different reference method, such as the determination of PWV by magnetic resonance imaging17. The great advantage of the new method is the ability to estimate PWV with a conventional BP cuff on the upper arm, regardless of the examiner, fully automatically and quickly and at affordable prices, and also in clinical settings such as community pharmacies.

Vascular age (VA) can be defined by age-adjusted percentiles of estimated PWV assessed with oscillometry, because estimated PWV shows a monotonous increase with age. The difference from expected estimated PWV, just based on chronological age, allows classification into normal, higher PWV or premature (or early) VA and lower PWV or healthy VA. In other words, higher VA means the estimated PWV is above the 90th percentile for the corresponding age group, lower VA means the estimated PWV is below the 10th percentile for the corresponding age group. Following this reasoning in arterial damage, the concept of "early vascular aging (EVA)" has been developed in recent years, i.e. accelerated vascular aging, suggesting that there is a difference between chronological age, defined by date of birth, and biological age, characterized by the actual state of the vascular tree. The expression "Your arteries are 10 years older than you" in a hypertensive patient with increased arterial stiffness, aims to make one understand that the arteries have aged prematurely by the action of risk factors on a given genetic background. The same reasoning is used to express the VA of patients according to the intima-media thickness in the carotid bed. Arterial wall alterations measured in practice can therefore be translated into concepts such as arterial aging and VA.

The predictive value of HMOD represents a complementary and additional concept to traditional risk tables. The risk tables remain valid and should be the first instrument applied to all patients to establish their CV risk. The peculiarity of HMODs is that they improve risk stratification beyond the tables. Sehestedt demonstrated already in 2010 in a pioneering study conducted in approx. 2,000 subjects without previous CV disease, which included adjusting for the SCORE tables, that the greater the number of HMODs, the greater the risk of patients suffering a CV event in the following 12 years. Studies carried out in our environment by researchers participating in TOGETHER, such as the MARK Study, confirm the relevance of arterial stiffness as an instrument for improving the stratification of CV risk in subjects initially classified as medium risk. 2,449 participants were recruited in 6 primary care centers in 3 Autonomous Communities, with a prevalence of vascular damage of up to 44%.

This last aspect, although in a cross-sectional design, has been studied recently in 923 people who entered community pharmacies in the Valencian Community, who were offered to determine their CV risk based on SCORE. Almost 51% of participants could not classify their CV risk either because they were below 40 years or above 65 years; thus, did not fall into the applicable age limits for SCORE. In this group, however, ePWV over the 90th percentile of the corresponding age-group were diagnosed in 18% of cases. In the remaining half, susceptible to evaluation by SCORE, only 2% presented with high or very high vascular risk according to the SCORE tables, while ePWV from brachial oscillometry, and therefore HMOD and elevated risk, were present in almost 10% of participants, that is, with a frequency five times higher. There are abundant examples in the literature that the detection of HMOD contributes to correctly reclassifying the CV risk of patients, also in other organs.

In summary, by estimating arterial stiffness through brachial oscillometry it may be possible to diagnose subclinical arterial damage, translated into the concept of VA and accelerated arterial aging, thus improving risk stratification.

Difficulties in understanding the traditional concept of "cardiovascular risk" Classical risk factors such as HTN, dyslipidemia and smoking are characterized by the lack of symptoms, and therefore do not generate the need for patients to consult their doctor for symptomatic reasons. We have previously noted that risk tables significantly improved risk stratification by merging into a single variable the damage produced by five established CV risk factors. However, it represents a theoretical concept that is generally outside the scope of understanding of most citizens. According to the most recent SCORE2 reference tables, the CV risk unit shown in the tables corresponds to the risk of suffering a fatal or non-fatal CV event within 10 years of the determination. This definition, to be explained to a layperson in medicine, implies understanding what is a fatal and non-fatal CV event, as well as realization that probabilities of events, expressed in percentages, are being estimated in a time frame of 10 years. Transmitting that knowledge is certainly possible, but it is not simple and takes time.

Arterial stiffness, estimated as PWV (ePWV) by brachial oscillometry, offers a simpler alternative. Based on a reference group of more than 1,900 people and with a wide age distribution, between 14 and 99 years, a study was carried out that defined specific ePWV reference values for seven age groups in terms of percentiles20. These reference values have recently been evaluated in the Heinz Nixdorf Recall Study, a population study in the Ruhr area in Germany. As a result, it is now possible to calculate for each subject individually, if the measured VA value is below the 50th percentile, between the 50th and 90th percentile, or above the 90th percentile. A simple graphic representation in the form of the system of traffic lights (red-yellow-green) serves for the patient to understand the measured value and obtain a direct visual reference on what is the state of his arterial system and his VA estimated by a single image, similar to the risk associated with food intake based on its fat content in some European countries. The TOGETHER Project will assume the same visual alert system to translate medical pathophysiological variables simply and directly into messages understandable to patients.

In the study "Measuring vascular age in Upper Austria", a feasibility study was carried out to determine whether it is possible to register BP and VA on a large scale in community pharmacies at the same time. Over a period of about one and a half years, BP and VA were measured with a special BP cuff ("AGEDIO®, IEM, Stolberg, Germany) at 45 public pharmacies and at 2 health events in Upper AT. Despite a cost of 10 Euros for patients, the offer to perform a measurement was accepted by more than 10,000 people. Overall, 37.3% were above the 90th reference percentile (EVA), with proportions rising from one-quarter in youngest to one-half in oldest participants.

Similar feasibility studies have also been conducted in Spain and Portugal to validate estimating VA in community pharmacies. In the RIVALFAR study, carried out in the Valencian Community, community pharmacies determined ePWV with the same device (AGEDIO®, IEM, Stolberg, Germany) in 1,427 subjects who entered those pharmacies. An elevated arterial stiffness frequency of 28.4% of the participants was recorded, and it was found that the determinants of this stiffness coincided with those described in the literature on EVA, i.e., male gender, age, pulse pressure, abdominal obesity and heart rate, thus demonstrating the ability of properly trained community pharmacies to measure arterial stiffness and transmit results to patients. Finally, the ASINPHAR@2action project also confirmed in Portugal the suitability and capacity of community pharmacies to estimate vascular age with brachial oscillometry, using the same device (AGEDIO®, IEM, Stolberg, Germany). The frequency of increased arterial stiffness in the 658 participating subjects was 19.8%. Factors predicting presence of pathological arterial stiffness were age, gender, aortic PP, visceral fat, HDL cholesterol, Augmentation Index, total vascular resistance, HTN, and diabetes, also in line with the known determinants of VA. It is important to underline that all three studies, "Measuring vascular age in Upper Austria", the "RIVALFAR study" and the "ASINPHAR@2action project" were carried out independently from each other.

Deficiencies in structured health education of hypertensive subjects In this context, it is essential to refer to patient health education as one of the most important pillars for improving BP control. There is enough evidence in the literature to say that health education represents an effective measure to control HTN, regardless of whether it is carried out in health centers, medical consultations or community pharmacies . One recent study confirmed that motivating patients to adopt healthier lifestyles and improve CV risk profile by communicating their Heart-Age, according to the so-called "Heart-Age tool", was superior to the traditional percentage-based tables. Overall, 3,153 patients were randomly allocated to firstly, either the control group, based exclusively on conventional medical advice, or secondly, to the Framingham REGICOR, a 10-year percentage risk score, calibrated to Spanish population or thirdly, the Heart Age group, where the concept of Heart Age was explained to the subjects. The latter group significantly reduced the CV risk after one year compared to the other groups, suggesting that the use of simple concepts, such as heart age opposed to chronological age, improved risk perception in the general population.

Bakhit et al published recently a meta-analysis including 62 randomized trials that compared any CV disease risk communication strategy versus usual care in terms of accuracy of risk perception, clinician-reported changes in CV risk, psychological responses, intention to modify lifestyle, self-reported changes in risk factors and clinician prescribing of preventive medicine. It could be shown that any kind of risk communication led to a small but significant BP reduction, mainly by improvement of the CV risk perception and increase in medication adherence.

At the international level, many studies have demonstrated the relevant role of the community pharmacist in the primary and secondary prevention of CV. A study of 56 randomly selected community pharmacies found a significant reduction in systolic BP, LDL cholesterol and CV risk (21%) in the group of patients who had received adequate counseling and follow-up in pharmacies. Evidence from systematic reviews with meta-analyses supports that pharmacist interventions, alone or in collaboration with other healthcare professionals, improve BP management. However, the effect of these interventions is heterogeneous.

In addition, interventions by the community pharmacist have been shown to be the most effective for the patient: interventions focused on the control of HTN and diabetes, followed by total and LDL cholesterol control. Many of these interventions included monthly follow-up focused on adherence to nutritional guidelines and modification of lifestyle habits (physical exercise and smoking cessation), as well as patient education and counseling about lifestyle, feedback to physicians, medication adherence and medication management. Moreover, recent guidelines on HTN, notably the 2017 guidelines from the American College of Cardiology and the American Heart Association as well as the 2023 guidelines of the ESH recommend the involvement of pharmacists for the team-based management of HTN.

Absence of structured communication between Primary Care Physicians and Community Pharmacies GPs and Community Pharmacists represent two key actors in the management of all health care systems, regardless of their structural diversities. Several initiatives document the willingness of collaboration between both groups, specifically in the field of HTN. Thus, in ES, consensus guidelines have been published regarding the referral of hypertensive patients from the pharmacy to the GPs and the role of pharmacists in HTN. Joint training programs in HTN (IMPACHTA) have been developed, however, there are no public or private programs integrating these two actors of health systems in an institutional way, especially not for the control of specific pathologies, such as HTN.

In a survey including 212 GPs throughout Spain (MAPHA), only 14% of hypertensive patients were diagnosed in collaboration with community pharmacies. In the same survey, 26.2% of GPs stated that they had no relationship with pharmacists in their environment, and 13.8% expressed a lack of confidence in their measures. However, 60.0% of the respondents were satisfied that pharmacists were responsible for monitoring the BP of their HTN patients. The literature has described validated surveys that analyze the relationship between pharmacists and GPs, but their implementation is limited to the scope of research and do not yet form part of daily clinical and pharmaceutical practice.

The objective of this study is to develop collaborative programs aimed at lightening the burden of primary care, improving health education shared between community pharmacies and GPs, whether in health centers or private consultations, and to improve both the early diagnosis of HTN and its control.

Design This protocol is based on the hypothesis that the concept of "Vascular Age", being more accessible and easy to grasp than other medical terms, will help hypertensive patients to better understand their CV risk. Our hypothesis assumes that this awareness of the state of their health will empower them to take actions in pursuit of its improvement, resulting in a better interaction with health care providers as well as in a better control of their BP compared to patients who received the usual medical care.

Likewise, we think that the empowerment of patients through knowledge of their VA will establish a link of greater trust between GPs and the Community Pharmacies participating in the study, compared to the usual care. The TOGETHER Project has a longitudinal cluster-randomized prospective design with two cohorts:

* BP Cohort: This is the usual care cohort. At baseline visit BP will be measured, followed by usual care. ePWV will be also determined in a blinded fashion (for comparison of the baseline variables), but it will not be communicated neither to the pharmacist or the GP, nor to the patient, till the end of the study.
* EVA Cohort: As in the BP cohort, BP will be measured at baseline, and in addition, ePWV from brachial oscillometry will be assessed to determine VA, which will be communicated to the patient, the pharmacist and the GP.

After stratification by region, each participating community pharmacy will be assigned a cohort type randomly, providing a homogeneous geographical distribution so that ~50% of pharmacies will communicate only BP (BP cohort) and 50% will communicate BP and vascular age (EVA cohort), using the strategy of cluster randomization. No inclusion number per pharmacy is set a priori. The number of patient inclusions is monitored country-specifically. After the specified total number of participants in a country has been reached, the pharmacies are informed that the acquisition of study participants must be stopped. The expected recruitment time will be at least six months.

Primary and Secondary outcomes Given the main objective of evaluating the extent to which knowledge of VA improves the control of HTN, the following primary and secondary endpoints are defined.

Procedures All study procedures are in accordance with recent guidelines. Recruitment of Community Pharmacies takes place through previous collaborations and/or invitation from public institutions, either the Austrian Chamber of Pharmacists / Upper Austria (APO), or scientific societies such as SEFAC, Spanish Society of Family and Community Pharmacies in Spain. The random allocation of the Community Pharmacies to the BP cohort or the EVA cohort follows cluster-randomization, which takes place according to criteria of regional homogeneity.

Trained pharmacy personnel will measure BP in Community Pharmacies according to a standard procedure following the 2023 European Society of Hypertension Guidelines for the Management of Arterial Hypertension13, using automated attended triple measurement, and the BP shown is the average of the second and third measurement. In addition, the estimation of VA by brachial oscillometry with the same device, Tel-O-Graph® (IEM, Stolberg, Germany) will be performed in both the BP and the EVA cohort. In the BP cohort, this will be done in a blinded way, and the results will not be disclosed to patient, pharmacist or physician. In the EVA cohort, the results will be shown to the pharmacist, discussed with the patients and reported to the physician.

Participants presenting with BP ≥ 140 mmHg and/or diastolic BP ≥ 90 mmHg will be invited to participate in the study. If the individual agrees and after explaining the aims of the study, study procedures, advantages and disadvantages of participating, the informed consent (IC) will be signed and the individual will enter the study. Standardized education concerning HTN will then be given by trained pharmacy personnel in both cohorts (BP and EVA) in face-to-face meetings. In the EVA cohort, additional education about VA will be provided.

1. Austria:

   Patients in both cohorts receive the recommendation to see their family doctor for further work up and, eventually, treatment of the elevated BP. Pharmacies prepare a report for the family doctor that contains the following:
   1. BP-cohort: the result of the BP measured in the pharmacy.
   2. EVA-cohort: the result of the BP measured in the pharmacy and VA. The GP performs ABPM, using the Mobil-O-Graph® device (IEM, Stollberg) to confirm elevated BP. If ABPM BP is not elevated (24-hour average SBP < 130 and DBP < 80 mm Hg), the patient will leave the study. If the BP is elevated, the GP will provide standardized BP education in both study cohorts. In addition, education is provided on the importance of VA and the prognostic consequences of increased VA in the EVA cohort. The education takes place in personal meetings or online by trained staff with the help of visual material that is adapted from ongoing BP training projects (herz.leben in Styria PharmaFit in Madrid and Team-Based Care (TBC-HTA) in Switzerland. The standardized education on VA in the EVA cohort takes place in personal meetings in small groups by trained staff in the GP´s office using visual material adapted from the European COST (European Cooperation in Science and Technology) Action VascAgeNet ("Network for Research in Vascular Ageing") . The Upper Austrian Society for General and Family Medicine (OBGAM) and the study advisor will carry out the training for specialized staff in GP offices.
2. Spain/Portugal:

After study inclusion and the first education about BP (both cohorts) or VA (EVA cohort only), ABPM is carried out in the pharmacies using the Mobil-O-Graph® device (IEM, Stollberg). If ABPM BP is not elevated (24-hour average SBP < 130 and DBP < 80 mm Hg), the patient will leave the study. If BP is elevated, standardized BP education will be provided in the health centers assigned to the pharmacies in both study cohorts. In addition, education is provided on the importance of VA and the prognostic consequences of increased VA in the EVA cohort. The education on BP and on VA will be standardized and identical to the training in AT. The scientific society SEMERGEN (Spanish Society of Primary Care Physicians) or the Primary Investigator will carry out the training for the specialist staff in the health centers. Pharmacies prepare a report for the family doctor that contains the following:

1. BP-cohort: the result of the BP measured in the pharmacy.
2. EVA-cohort: the result of the BP measured in the pharmacy and VA, the result of the laboratory measurement and the result of SCORE/SCORE2.

A determination of the most important CV risk markers (total cholesterol in ES/PT and total cholesterol, LDL, HDL cholesterol, triglycerides in AT) is carried out either in the pharmacy (ES/PT) or in the doctor´s office (AT) as part of clinical routine. This allows CV risk to be calculated according to the SCORE/SCORE2 tables.

In both ES/PT and AT, patients are managed and treated by the GP in accordance with the ESH 2023 HTN Guidelines and clinical experience. The GP can request further examinations that he/she considers appropriate and that are not part of the study, such as: e.g. resting ECG, echocardiogram etc.

A second ABPM will be performed between 3 and 6 months after the first ABPM, in ES/PT in the community pharmacies, in AT by the GP. At the same time as the second ABPM, the following measurements are also carried out in ES/PT and transmitted to the family doctors. BP-cohort: BP measured in the pharmacy, cholesterol levels and calculation of SCORE/SCORE2; EVA-cohort: BP measured in the pharmacy, cholesterol levels and calculation of SCORE/SCORE2. At the same time as the second ABPM, office BP is measured in AT by the GP. The study ends with the second ABPM. The patients are further treated by their GPs according to clinical routine. It is readily available to the family doctors in AT and will be sent to them in a report in ES/PT (see above).

At the beginning of the study, in all patients, pharmacists and GPs will complete validated questionnaires to evaluate the interaction between them, while patients will be given questionnaires to assess adherence. This will be repeated at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* BP ≥ 140 mmHg and/or ≥ 90 mmHg in the pharmacy
* 24-hour ABPM ≥ 130 mmHg or ≥ 80 mmHg
* Willingness to fill in forms, regarding

  * Anamnesis (DM, hypercholesterolemia)
  * Toxic habits
  * Pharmacological groups of CV medication
  * Previous CV diseases
  * Data on GP and assigned Health Center
  * Survey regarding interaction with GP and community pharmacist

Exclusion Criteria:

* Pregnancy
* Inability to understand the project (language barrier)
* Manifest incapacity or knowledge of the existence of a legal representative
* Factors preventing the correct measurement of BP/VA (arrhythmias, arm circumference, etc.)
* Previous measurement of VA in the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1246 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in the EVA cohort who do comply with the visit to the Primary Care Physician compared to the proportion of patients in the BP cohort who do comply with the visit to the Primary Care Physician. | Time between enrollment and diagnosis of hypertension in the community pharmacy and referral to the visit by the Primary Care Physician will be four weeks.
  Hypertensive patients will be randomized to the BP-cohort or the EVA-cohort. The hypothesis of the study is that the proportion of patients in the EVA-cohort who comply with the visit to the Primary Care Physician will be significantly higher than the proportion of patients in the BP-cohort who comply with the visit to the Primary Care Physician. Independent variables: Cohort [BP/EVA], Sex [f/m], Age [years], SBP [mmHg], DBP [mmHg], Smoker [yes/no], Heart rate [beats/min], Diabetes [yes/no], Obesity [yes/no], Pulse pressure (SBP - DBP) [mmHg], Prior CV event [yes/no].
  In case of normal distribution of continuous variables but lack of variance homoscedasticity, Welch's t-test will be applied. For comparisons of continuous variables without normally distributed data and for comparisons of variables measured on ordinal scales, the Mann-Whitney U-test will be used. Dichotomous variables will be compared by the Fisher´s exact test, all other categorical variables by the chi-square test.
Proportion of hypertensive patients in the EVA cohort who normalize blood pressure compared to the proportion of hypertensive patients in the BP cohort who normalize blood pressure as assessed by a second ABPM six months after the first ABPM. | Time between the first and the second ABPM will be six months
  Hypertensive patients will be randomized to the BP-cohort or the EVA-cohort. The hypothesis of the study is that patients in the EVA-cohort who normalize BP in the second ABPM will be significantly higher than the proportion of patients in the BP-cohort who normalize BP as assessed in the second ABPM. Normal ABPM means ABPM 24-h < 130/80 mmHg.
  Independent variables: Cohort [BP/EVA], Sex [f/m], Age [years], SBP [mmHg], DBP [mmHg], Smoker [yes/no], Heart rate [beats/min], Diabetes [yes/no], Obesity [yes/no], Pulse pressure (SBP - DBP) [mmHg], Prior CV event [yes/no].
  In case of normal distribution of continuous variables but lack of variance homoscedasticity, Welch's t-test will be applied. For comparisons of continuous variables without normally distributed data and for comparisons of variables measured on ordinal scales, the Mann-Whitney U-test will be used. Dichotomous variables will be compared by the Fisher´s exact test, all other categorical variables by the chi-square test.

SECONDARY OUTCOMES:
Change of 5 mmHg in systolic blood pressure and/or of 2 mmHg in diastolic blood pressure in the second ABPM | Six months between first and second ABPM.
  The proportion of patients in the EVA cohort with a change of 5 mmHg in systolic blood pressure and/or of 2 mmHg in diastolic blood pressure in the second ABPM will be significantly greater than in the BP cohort.
Changes in lipid metabolism of cholesterol-LDL towards normalization. | Six months.
  The proportion of patients in the EVA arm who will normalize their cholesterol-LDL will be significantly higher than the proportion of patients in the BP arm. The threshold for normal cholesterol-LDL is 115 mg/dl.
Change of body mass index (BMI) from obesity towards overweight or normal weight. | Six months.
  The proportion of patients in the EVA arm who will normalize their weight will be significantly higher than the proportion of patients in the BP arm. The threshold for normal weight, assessed as body mass index, is < 30 m/m2.
Change in proportion of smokers who quit smoking. | Six months.
  The proportion of patients in the EVA arm who will quit smoking will be significantly higher than the proportion of patients in the BP arm. The outcome is dichotomous (yes/no) and will be assessed by a asking directly those patients who were smokers at baseline.
Changes in vascular risk stratification. | Six months.
  The proportion of patients in the EVA arm who will achieve low or moderate cardiovascular risk according to SCORE2 will be significantly higher than the proportion of patients in the BP arm. The cardiovascular risk table used will be SCORE2, which describes four different CV risk groups: low (< 1%), moderate (1-4%), high (5-9%), very high (> 9%), the unit is the probability of suffering a CV event in the following ten years.
Changes in the score of collaborative surveys between Pharmacists and Primary Care Physicians. | Six months.
  Pharmacies will be randomized a priori into two groups, those who measure only Blood Pressure (BP) and those who measure Blood Pressure and Early Vascular Aging (EVA). The hypothesis of the study is that empowerment of hypertensive patients by knowledge of their EVA will increase their adherence to treatment and improve the collaboration and the success of treating hypertension between pharmacists and physicians. A validated questionnaire published by Zillich et al. (Utility of a questionnaire to measure physician-pharmacist collaborative relationships. J Am Pharm Assoc (2003). 2006 Jul-Aug;46(4):453-8. doi: 10.1331/154434506778073592.) measures the relationship between these groups. The questionnaire includes 13 questions, each scored 1-7, the higher the sum, the better the collaboration. The questionnaires will be performed at the beginning and at the end of the study. The hypothesis is that the score of collaboration will be significantly higher in the EVA cohort.
Change in scores measuring adherence with prescribed antihypertensive treatment. | Six months.
  Pharmacies will be randomized a priori into two groups, those who measure only Blood Pressure (BP) and those who measure Blood Pressure and Early Vascular Aging (EVA). The hypothesis of the study is that empowerment of hypertensive patients by knowledge of their EVA will increase their adherence to treatment and improve blood pressure control. A validated questionnaire published by Stone at al. (https://doi.org/10.1093/ibd/izaa056) estimates adherence to antihypertensive treatment. The questionnaire includes 5 questions, each scored 1-5, the higher the sum, the better the adherence. The questionnaires will be performed at the beginning and at the end of the study. The hypothesis is that adherence will be significantly better in the EVA cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Weber, PhD, full Professor, Study Chair — Cardiology Department, Klinikum Wels-Grieskirchen, Wels, Austria
Locations (6):
- Austria (2):
  - Austrian Chamber of Pharmacists, Upper Austria (APO), Linz
  - Upper Austrian Society for General and Family Medicine (OBGAM), Linz
- H&TRC - Health & Technology Research Center, Coimbra Health School, Polytechnic University of Coimbra, Coimbra, Portugal
- Spain (3):
  - Hospital de Sagunto, Sagunto (valencia), Valencia
  - Instituto Pluridisciplinar, Universidad Complutense de Madrid, Madrid
  - Unidad de investigación de Atención Primaria de Salamanca (APISAL). Instituto de Investigación Biomédica de Salamanca (IBSAL), Salamanca

IPD SHARING:
Plan to Share IPD: Yes
Due to the sensitive nature of the data (health data, medication prescription and adherence), it will be made available under a closed license according to which applicants will have to submit a proposal mentioning their goals and methodology to be granted access to the data and permission to reuse it. A data sharing agreement between the external party and the investigator will need to be agreed on and signed.
Supporting Information: Study Protocol, CSR
Time Frame: 01/JAN/2027 - 01/JAN/2028
Access Criteria: Applicants will have to submit a proposal mentioning their goals and methodology to be granted access to the data and permission to reuse it. A data sharing agreement between the external party and the investigator will need to be agreed on and signed.

REFERENCES:
- [Background] Danninger K, Hafez A, Binder RK, Aichberger M, Hametner B, Wassertheurer S, Weber T. High prevalence of hypertension and early vascular aging: a screening program in pharmacies in Upper Austria. J Hum Hypertens. 2020 Apr;34(4):326-334. doi: 10.1038/s41371-019-0222-y. Epub 2019 Jul 29. PMID 31358883
- [Background] Pereira T, Paulino E, Maximiano S, Rosa M, Pinto AL, Mendes MJ, Brito J, Soares P, Risse J, Gose S. Measurement of arterial stiffness and vascular aging in community pharmacies-The ASINPHAR@2action project. J Clin Hypertens (Greenwich). 2019 Jun;21(6):813-821. doi: 10.1111/jch.13554. Epub 2019 May 16. PMID 31095865
- [Background] Rodilla Sala E, Adell Alegre M, Giner Galvan V, Perseguer Torregrosa Z, Pascual Izuel JM, Climent Catala MT; en nombre del Grupo de estudio RIVALFAR. Arterial stiffness in normotensive and hypertensive subjects: Frequency in community pharmacies. Med Clin (Barc). 2017 Dec 7;149(11):469-476. doi: 10.1016/j.medcli.2017.04.037. Epub 2017 Jul 12. English, Spanish. PMID 28709670
- [Background] Rodilla E, Adell M, Baixauli V, Bellver O, Castillo L, Centelles S, Hernandez R, Martinez S, Perseguer Z, Prats R, Ruiz D, Salar L, Climent M; COPHARTEN Study Group. Value of estimating pulse wave velocity compared to SCORE in cardiovascular risk stratification in community pharmacies. Med Clin (Barc). 2023 Dec 7;161(11):463-469. doi: 10.1016/j.medcli.2023.06.002. Epub 2023 Sep 19. English, Spanish. PMID 37735046